CLINICAL TRIAL: NCT07299149
Title: A Prospective, Open-label, Single-arm Multicenter Clinical Study of Zanubrutinib, Obinutuzumab, and Lenalidomide (ZGR) in the Treatment of Untreated Follicular Lymphoma
Brief Title: Zanubrutinib, Obinutuzumab Combined With Lenalidomide (ZGR) for the Treatment of Untreated Follicular Lymphoma
Acronym: ZGR in TN FL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025107
Record Dates: First submitted 2025-11-21; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; zanubrutinib; Obinutuzumab; lenalidomide
MeSH Terms: conditions — Lymphoma, Follicular | interventions — obinutuzumab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Induction therapy of ZGR, and maintenance therapy of ZR (Experimental): Induction therapy: All enrolled patients received the ZGR regimen (zanubrutinib, obinutuzumab, and lenalidomide) for Cycles 1-4. Tumor response was assessed after Cycle 4. Patients achieving complete response (CR) or partial response (PR) continued the same ZGR regimen for 2 additional cycles (Cycles 5-6).
  Maintenance therapy: After completing induction therapy, patients with sustained CR/PR initiated maintenance therapy with zanubrutinib plus lenalidomide (ZR) for 18 months (1.5 years) or until disease progression, intolerable toxicity, or trial withdrawal (whichever occurred first)
  Interventions: Drug: Induction Therapy: Zanubrutinib, obinutuzumab, lenalidomide; Drug: Maintenance therapy: Zanubrutinib, lenalidomide

INTERVENTIONS:
Drug: Induction Therapy: Zanubrutinib, obinutuzumab, lenalidomide — All enrolled patients received: Zanubrutinib: 160 mg twice daily, orally, on Days 1-28; Obinutuzumab: 1000 mg, intravenous infusion: Days 1, 8, and 15 of Cycle 1,on Day 1 of Cycles 2-6; Lenalidomide: 25 mg once daily, orally, on Days 1-21 of each 28-day cycle.
Drug: Maintenance therapy: Zanubrutinib, lenalidomide — Maintenance therapy consists of zanubrutinib plus lenalidomide: Zanubrutinib: 160 mg twice daily, orally, on Days 1-28.Lenalidomide: 25 mg every other day, orally, on Days 1-21 of each 28-day cycle

SUMMARY:
This study is planned to prospectively evaluates the efficacy and safety of the zanubrutinib, obinutuzumab, and lenalidomide (ZGR) combination regimen in treatment-naïve follicular lymphoma (FL) patients in a Chinese population.

DETAILED DESCRIPTION:
Regarding chemotherapy-free first-line treatment regimens, current targeted therapies primarily focus on lenalidomide combined with anti-CD20 antibodies. Chemotherapy-free regimens such as rituximab plus lenalidomide (R²) or obinutuzumab plus lenalidomide (O-Len) have been recommended for clinical use. Encouraged by the promising efficacy of dual-targeted therapies, the potential of triple-combination therapy-comprising a BTK inhibitor (BTKi), an anti-CD20 monoclonal antibody, and lenalidomide-has garnered increasing attention in untreated hematologic malignancies. Most existing studies have concentrated on BTKi combined with rituximab and lenalidomide (e.g., ibrutinib + R²).

Given current clinical needs and available evidence, this study aims to explore a novel chemotherapy-free triple regimen: zanubrutinib combined with obinutuzumab and lenalidomide (ZGR) in treatment-naïve follicular lymphoma (FL) patients. This combination is expected to provide a new treatment paradigm for untreated FL, offering high antitumor efficacy while minimizing toxicity, thereby improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Gender: No restrictions; age ≥18 years.
* Diagnosis: Histologically confirmed CD20-positive follicular lymphoma (FL), Grade 1, 2, or 3A, per 2016 WHO classification. All patients must provide sufficient archived or fresh tumor tissue samples for immunohistochemical (IHC) analysis.
* Disease Stage & Treatment Need:
* Stage III or IV disease, or Stage II with bulky disease, meeting at least one of the following criteria:
* a) Bulky disease: Lymph node or extranodal (excluding spleen) mass with maximum diameter ≥7 cm.
* b) Local symptoms or organ dysfunction due to progressive lymphadenopathy or extranodal tumor mass.
* c) B symptoms (fever, night sweats, or unintentional weight loss >10% of body weight within ≤6 months).
* d) Symptomatic extranodal involvement (e.g., pleural/peritoneal effusion).
* e) Cytopenias due to bone marrow infiltration (hemoglobin <10 g/dL, absolute neutrophil count [ANC] <1.0×10⁹/L, platelets <100×10⁹/L).
* f) Involvement of ≥3 lymph nodes, each ≥3 cm in diameter.
* g) Symptomatic splenomegaly.
* Prior Therapy: No prior systemic therapy for FL.
* ECOG Performance Status: ≤2.
* Measurable Disease: At least one measurable lesion (>2 cm in longest diameter by CT/MRI).
* Life Expectancy: ≥6 months.
* Adequate Organ Function:
* a) ANC ≥1.0×10⁹/L (without growth factor support).
* b) Platelets ≥50×10⁹/L (untransfused within 7 days).
* c) Total bilirubin (TBIL) ≤1.5×ULN.
* d) ALT/AST ≤3×ULN.
* e) Creatinine clearance ≥30 mL/min (calculated by modified Cockcroft-Gault formula).
* Contraception: Men and women of childbearing potential must agree to use highly effective contraception during the study and for 4 weeks after treatment discontinuation.
* Informed Consent: Patients must voluntarily participate and sign informed consent forms (ICF).

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from this study:
* Histologic evidence of central nervous system (CNS) lymphoma, leptomeningeal lymphoma, or transformation to high-grade lymphoma (e.g., diffuse large B-cell lymphoma, DLBCL).
* Grade 3B follicular lymphoma (FL) or transformed FL.
* Ann Arbor Stage I FL.
* Prior history of malignancy, unless the patient has been disease-free for ≥5 years and the treating physician deems the risk of recurrence low (exceptions: non-melanoma skin cancer, cured localized prostate cancer, carcinoma in situ of the cervix, or squamous intraepithelial lesions on PAP smear).
* Use of any investigational drugs, antibiotics, or participation in another interventional clinical trial within 4 weeks prior to enrollment.
* Major surgery (excluding lymph node biopsy) within 14 days before enrollment or anticipated need for major surgery during the study.
* Prior treatment with zanubrutinib, obinutuzumab, or lenalidomide.
* Immunodeficiency or autoimmune disease history, or chronic systemic steroid therapy (>10 mg/day prednisone equivalent) or immunosuppressive therapy within 7 days before enrollment.
* Severe hepatic dysfunction (including severe jaundice, hepatic encephalopathy, refractory ascites, or hepatorenal syndrome), cachexia, or multi-organ failure with renal impairment.
* Clinically significant cardiovascular abnormalities:
* NYHA Class III/IV heart failure
* Myocardial infarction within 6 months before enrollment, Malignant arrhythmias (including QTc ≥480 ms), Uncontrolled hypertension (Systolic blood pressure (SBP) ≥150 mmHg and diastolic blood pressure (DBP) ≥100 mmHg), Unstable angina.

Active infections:

* HIV, active hepatitis B/C infection (HBV DNA ≥2000 IU/mL or HCV RNA detectable)
* Uncontrolled systemic infections.
* Bleeding disorders or coagulation abnormalities, or thrombotic events within 3 months.
* Severe hypersensitivity to the active ingredients or excipients of the study drugs.
* Pregnancy, lactation, or unwillingness to use effective contraception in women of childbearing potential.
* Other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-04-28 (Estimated); Study Completion 2030-12-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate，ORR | up to the end of 6 cycles of treatment(each cycle is 28 days)]
  Defined as the proportion of patients with complete or partial response as assessed by response to induction therapy

SECONDARY OUTCOMES:
Complete response rate，CRR | up to the end of 6 cycles of treatment(each cycle is 28 days)
  defined as the proportion of patients with complete response as assessed by response to induction therapy.
Best overall response rate (ORR) and complete response rate (CRR) during treatment | Up to the end of 6 cycles of treatment(each cycle is 28 days)
  defined as the proportion of patients with best response as assessed in the induction therapy.
CRR and ORR at end of treatment | at the end of Cycle 24 (each cycle is 28 days)
  Defined as the proportion of patients with complete response, and complete or partial response as assessed by response to the end of treatment(induction + maintenance therapy)
Progression-free survival (PFS) | up to 5 years
  The time from the enrollment of a subject to the occurrence of (in any way) progression of disease or Death for any reason. patients with indeterminate recurrence or Death at the last follow-up, defined as the date of the last Investigation
Duration of response (DOR) | up to 5 years
  defined as the time from the first treatment response (including complete response and partial response) to the last assessment of response.
Time to response (TTR) | at the end of Cycle 24 (each cycle is 28 days)
2-year overall survival (OS) rate | up to 2 years
  The time from subject enrollment to Death caused by any reason. for patients lost to follow-up, the time of the last follow-up; for patients still alive at the end of study, the date of the end of follow-up
Proportion of patients with progression of disease within 24 months (POD24) | Up to the end of 2 years (each cycle is 28 days)
The safety | up to 5 years
  Incidence of adverse events, serious adverse events and significant adverse event

OTHER OUTCOMES:
Minimal residual disease (MRD) monitoring | Up to the end of 24 cycles of treatment(each cycle is 28 days)
Circulating tumor DNA (ctDNA) analysis via next-generation sequencing (NGS) | Up to the end of 24 cycles of treatment(each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, Tianjin 300020, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No